CLINICAL TRIAL: NCT04692545
Title: Preoperative Immunonutrition Versus Standard Dietary Advice in Normo-nourished Patients Undergoing Fast-track Laparoscopic Colorectal Surgery
Brief Title: Preoperative Immunonutrition in Normonourished Patients Undergoing Fast-track Laparoscopic Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, MD, PhD, Associate Professor, University of Rome Tor Vergata
Other Study IDs: REGISTROSPERIMENTAZIONI /21
Record Dates: First submitted 2020-12-25; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immunonutrition Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: patients receiving immunonutrition supply
  Interventions: Dietary Supplement: Immunonutrition
- B: patients receiving standard dietary advice

INTERVENTIONS:
Dietary Supplement: Immunonutrition — nutridrinks 3 times a day 5 days prior surgery plus maltodextrins the day of surgery
  Groups: A

SUMMARY:
Immunonutrition (IN) appears to reduce infective complications and in-hospital length of stay (LOS) after gastrointestinal surgery. More specifically, it seems to be beneficial also in colorectal cancer surgery. Potential benefits of combining preoperative IN (PIN) with protocols of enhanced recovery after surgery (ERAS) in reducing LOS in laparoscopic surgery are yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic colorectal resection for cancer following ERAS protocol
* >18 years old
* elective setting

Exclusion Criteria:

* age below 18
* malnutrition
* inflammatory bowel disease
* acquired or congenital immunodeficiency
* preoperative infection
* ASA IV
* pregnancy
* emergency setting
* conversion to open surgery
* multivisceral resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All normonourished patients undergoing elective ERAS laparoscopic colorectal resections for cancer at Minimally Invasive Surgery Unit of Tor Vergata University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | up to 30 days after discharge
  number of days between primary colorectal resection and discharge

SECONDARY OUTCOMES:
Time to postoperative food intake | up to 30 days after discharge
  number of days between primary colorectal resection and refeeding
Time to first defecation | up to 30 days after discharge
  number of days between primary colorectal resection and first defecation
30-days postoperative complications | up to 30 days after discharge
  Rate of any complication after colorectal resection
Surgical site infection | up to 30 days after discharge
  rate of any surgical site infection clinically demonstrated
Anastomotic leak | up to 30 days after discharge
  rate of any postoperative leakage of colo-rectal, colo-colic or ileo-colic anastomosis, clinically, radiologically or endoscopically demonstrated
Readmission | up to 90 days after discharge
  Rate of any unplanned readmission after discharge
30-days Mortality | up to 30 days after discharge
  Rate of any mortality
Pneumonia | up to 30 days after discharge
  rate of radiologically demonstrated pneumonia
Ileus | up to 30 days after discharge
  rate of any ileus clinically demonstrated
Prolonged length of stay | up to 30 days after discharge
  rate of any patient discharged after 8 days

IPD SHARING:
Plan to Share IPD: No